CLINICAL TRIAL: NCT05693740
Title: Pulsed Light Versus Continuous Light Accelerated Epithelium-Off Cross-linking for Treatment of Progressive Keratoconus; a Prospective Comparative Study
Brief Title: Accelerated Corneal Collagen Crosslinking Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdel-Radi, Assistant professor Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: accelerated cross-linking
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Intervention Model Description: Single blinded Prospective, Interventional, randomized, comparative study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- group 1 (Active Comparator): Patients in this group will undergo pulsed light accelerated crosslinking (pl-ACXL)
  Interventions: Procedure: Accelerated crosslinking (ACXL)
- group 2 (Active Comparator): Patients in this group will undergo continuous-light accelerated crosslinking (cl-ACXL)
  Interventions: Procedure: Accelerated crosslinking (ACXL)

INTERVENTIONS:
Procedure: Accelerated crosslinking (ACXL) — Epithelium-off accelerated corneal crosslinking is a procedure in which the cornea is soaked with riboflavin followed by exposure to ultraviolet irradiation in either pulsed-light or continuous-light modes to strengthen the corneal stroma and halt keratoconus progression.

SUMMARY:
To evaluate and compare the effect of pulsed light (pl-ACXL) accelerated and continuous light accelerated (cl-ACXL) epithelium-off cross-linking in halting the progression of keratoconus.

DETAILED DESCRIPTION:
Keratoconus (KC), which was first described in detail in 1854, is the most common corneal primary ectasia and is characterized by progressive bilateral and asymmetric corneal thinning and bulging outward into a cone-like shape that can severely impact patients' vision.

Keratoconus usually develops in the second and third decades of life and progresses until the fourth decade. It was thought to be a rare corneal disease.

Despite a great deal of research, no one theory explains it all and it may be caused by a combination of things. However, Meek proposed that the loss of structural integrity in the KC cornea was caused by the presence of abnormal keratocytes and matrix proteins and upregulated proteolysis triggered an unravelling of lamellae along their length and from their anchors at the limbus, with an opening of the lamellar bifurcations. This theory is supported by observations following riboflavin/UVA collagen cross-linking, where the proposed cross-linkage of the tissue increases both the resistance of the stroma to enzymatic digestion and the cohesiveness between collagen fibrils and the non-collagenous matrix.

Conventional CXL (CXL) with a continuous irradiation of 3 mW/cm2 for 30 min is considered safe and effective in the prevention of keratoconus progression according to different clinical trials. nevertheless, the procedure is time-consuming, lasting around 1 h, which may lead to patient discomfort and reduced physician working efficiency.

With evolving technical advances, commercially available UV light sources have been developed, making CXL more efficient with shorter UV exposure times, higher UV intensities, and pulsed light compared with continuous light settings. Various accelerated CXL protocols have been described and its effect on biomechanical properties on corneas stated as equal to the standard protocol. Ex-vivo studies also suggest a distinction between various accelerated CXL protocols by providing evidence for a drop in efficiency with increased UV illumination intensity while maintaining equal surface energy. In this study we evaluate the two types of "accelerated crosslinking".

ELIGIBILITY:
Inclusion Criteria:

1. Patients with mild to moderate progressive keratoconus with maximum keratometry value Kmax < 56.0 D, Corneal thinnest pachymetry ≥ 400 µm and Corrected distance visual acuity (CDVA) equal to or better than 20/200 Snellen's acuity.
2. Established keratoconus progression:

   Increase of 1.0D or more in the manifest cylinder Increase of 0.5D or more in the manifest refraction spherical equivalent Increase of 1.0D or more in Kmax Increase of 0.75D or more in Kmean decrease of 2% or more in central thickness
3. Age: 18-40 y
4. Clear cornea

Exclusion Criteria:

1. Corneal scarring
2. Previous corneal surgery
3. Severe keratoconus wit non measurable refraction or Kmax ≥ 56 D or Corneal thinnest pachymetry < 400 µm

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
1. Visual outcome measures | one year following surgery
  Uncorrected and corrected distance visual acuity (UDVA & CDVA) using Snellen acuity chart
2. Refractive outcome measures | one year following surgery
  Manifest refraction spherical equivalent (MRSE) using Topcon autorefractometer
3. Topographic outcome measures | one year following surgery
  Scheimflug imaging device (Pentacam) for Diagnosis and follow up of Keratoconus after ACXL
Demarcation line depth | 3 months following surgery
  Demarcation line depth is an outcome used to assess the success of CXL procedure using anterior segment ocular coherence tomography (AS-OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Abdel-Radi, MD, Principal Investigator — Assiut University
Locations (1):
- Tiba eye center, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu Y, Reinach PS, Zhu H, Li L, Yang F, Qu J, Chen W. Continuous-light versus pulsed-light accelerated corneal crosslinking with ultraviolet-A and riboflavin. J Cataract Refract Surg. 2018 Mar;44(3):382-389. doi: 10.1016/j.jcrs.2017.12.028. PMID 29703291